CLINICAL TRIAL: NCT05658536
Title: The COPE Study: Pilot Intervention to Improve Symptom Self-management and Coping in Adults With Post COVID
Brief Title: The COPE Study: Pilot Intervention to Improve Symptom Self-management and Coping in Adults With Post COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Tracy Herring, Acting Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016345
Record Dates: First submitted 2022-12-16; First posted 2022-12-20 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Post COVID-19 Condition; Post-COVID-19 Syndrome
Keywords: Post-COVID-19; Self-management
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: A randomized, 2-group parallel design, 50-subject pilot clinical trial to examine the feasibility, acceptability, and initial effects of a telemedicine group-based intervention designed to improve symptom management and coping in adults with Post-COVID.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-Week Self-Management Group (Active Comparator): 6-week telemedicine group-based intervention designed to improve symptom management and coping in adults with Post-COVID. The intervention consists of six weekly group sessions that are 1.5 hours long. Group size is 8-10 participants.
  Interventions: Behavioral: 6-Week Self-Management Group
- 6-Week Waitlist Group (No Intervention): 6-week waitlist period during which participants will complete study assessments. After completing the study, waitlist participants will be offered the active intervention.

INTERVENTIONS:
Behavioral: 6-Week Self-Management Group — The goal of the 6-session group-based intervention for patients with Post-COVID is to teach patients behavioral strategies known to be helpful in managing several common Post-COVID symptoms, including fatigue, memory and attention issues, poor sleep, breathlessness, coping with anxiety and uncertainty, and stress management. It is currently available to patients who are seen in the Post-COVID-19 Rehabilitation and Recovery Clinic at UW and the Post-COVID-19 Clinic in VAPSHCS Rehabilitation Care Services.
  Arms: 6-Week Self-Management Group

SUMMARY:
This project is a randomized controlled pilot trial using mixed methods to examine the feasibility, acceptability, and initial effects of a telemedicine group-based intervention designed to improve symptom management and coping in adults with Post-COVID.

DETAILED DESCRIPTION:
Post-acute sequelae SARS-CoV-2 infection (PASC), also referred to as Post-COVID, is an emerging condition with debilitating symptoms relevant to rehabilitation medicine. Post-COVID has been described as the "next national health disaster". The Centers for Disease Control and Prevention describe Post COVID as a wide range of physical and mental health symptoms lasting four or more weeks after SARS-CoV-2 infection. Some of the most common and disabling symptoms include, fatigue, memory issues, pain-related symptoms, insomnia, and shortness of breath. In addition to these physical symptoms, many patients with Post-COVID report co-occurring mental health concerns, including anxiety and depression. It is believed that over 100 million people worldwide currently experience or have experienced Post COVID. Importantly, this condition can be debilitating and disabling - nearly one in five people reported not working as a direct result of Post COVID.

Psychosocial self-management interventions are a promising treatment for helping people with Post COVID manage their symptoms and engage in adaptive coping. Unfortunately, there is currently no cure for Post COVID, and it is unclear at what timepoint patients will recover or what proportion of patients will recover. Given the variability and chronicity of Post COVID symptoms, self-management interventions could be particularly beneficial. Research on patient populations with similar symptom profiles as Post COVID (e.g., myalgic encephalomyelitis, multiple sclerosis) suggests that psychosocial interventions like self-management can reduce symptom severity and interference and improve coping.

This randomized controlled pilot trial will use quantitative and qualitative methods to examine the feasibility, acceptability, and initial effects of a telemedicine group-based intervention designed to improve symptom management and coping in adults with Post-COVID.

The study objectives include:

1. To examine the feasibility and acceptability of a telemedicine group-based intervention for improving symptom management and coping in adults with Post-COVID.
2. To examine initial effects of a telemedicine group-based intervention on Post-COVID symptom management and adaptive coping.
3. To understand intervention participants' perceptions of the feasibility, acceptability, appropriateness, and perceived effectiveness of the Post-COVID intervention and their recommendations for improving the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Resident of Washington state
3. Diagnosis of a Post-COVID condition
4. Able to read, speak, and understand English
5. Availability of a telephone and internet access

Exclusion Criteria:

1. Severe cognitive impairment
2. Currently receiving other psychosocial treatments primarily for any Post-COVID symptom(s) or problem(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability | Collected via online survey at post-treatment (up to 2 months after Tx Session 6)
  Intervention Acceptability will be measured with the Acceptability of Intervention Measure (AIM). When assessed via online survey, responses from the Intervention Acceptability items will be averaged to create an average score [1-5]. A higher score indicates more agreement with intervention acceptability while a lower score indicates less agreement with intervention acceptability.
Intervention Appropriateness | Collected via online survey at post-treatment (up to 2 months after Tx Session 6)
  Intervention Appropriateness will be measured with the Intervention Appropriateness Measure (IAM). When assessed via online survey, responses from the Intervention Appropriateness items will be averaged to create an average score [1-5]. A higher score indicates more agreement with intervention appropriateness while a lower score indicates less agreement with intervention appropriateness.
Intervention Feasibility | Collected via online survey at post-treatment (up to 2 months after Tx Session 6)
  Intervention Feasibility will be measured with the Feasibility of Intervention Measure (FIM). When assessed via online survey, responses from the Intervention Feasibility items will be averaged to create an average score [1-5]. A higher score indicates more agreement with intervention feasibility while a lower score indicates less agreement with intervention feasibility.

SECONDARY OUTCOMES:
Depressive Symptoms | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Mood will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 8b. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of depressive symptoms.
Anxiety Symptoms | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Anxiety will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form 8a. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of anxiety.
Fatigue | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Fatigue will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 8a. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of fatigue.
Sleep Disturbance | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Sleep Disturbance will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 8a. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of sleep disturbance.
Perceived Cognitive Difficulties | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Perceived Cognitive Difficulties will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function - Abilities Short Form 8a. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of perceived cognitive difficulties.
Self-Efficacy | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Self-Efficacy will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions - Managing Symptoms Short Form 8a. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of self-efficacy.
Psychosocial Functioning | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Psychosocial Functioning will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities Short Form 8a. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of ability to participate in social roles and activities.
Pain Interference | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Change in Pain Interference will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 8a. When assessed via online survey, responses will be summed to form a total T-score score based on normative data. Higher scores indicate higher self-reported levels of pain interference.
Impression of Change | Collected via online survey at post-treatment (up to 2 months after Tx Session 6)
  Impression of Change will be measured with the Patient Global Impression of Change scale. Higher scores on this one-item scale indicate higher self-reported levels of impression of change.
Symptoms and Impact of Post-COVID | Collected via online survey at pre-treatment (up to 1 month before Tx Session 1) and post-treatment (up to 2 months after Tx Session 6)
  Symptoms and Impact of Post-COVID will be measured with the Long COVID Symptom and Impact Tools (ST and IT). When assessed via online survey, responses from the Long COVID Symptom Tool (ST) items will be scored as a simple count (yes/no). Higher scores indicate higher self-reported levels of symptoms of Post-COVID. Responses from the Long COVID Impact Tool (IT) will be summed. Higher scores indicate higher self-reported levels of impact of Post-COVID.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Herring, PhD, Principal Investigator — University of Washington; Lindsey Knowles, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Ninth and Jefferson Building, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make available to interested researchers a data file containing de-identified data used for each published article at the time the article is accepted for publication. The data will be de-identified to remove any variables from which it would be possible to identify any individual participants. Specifically, we will create a data file that includes all variables used in the published article and a list of the variables in the data file (along with variable labels) and send to investigators who request the data a copy of: (1) the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) the dataset (as an SPSS.sav file). Note, though, even though any data files that we share will be stripped of identifiers prior to release for sharing, it remains possible those who access the data could potentially use deduction to identify participants with unusual characteristics or combinations of unusual characteristics.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data used for the analyses for any papers published will become available to interested researchers by request after that article is published. Those data will continue to be available for at least five years following the publication of the article.
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Knowles LM, Grewal M, Drever SA, Hoffman JM, Friedly JL, Herring TE. A pilot randomized controlled trial of a telemedicine psychosocial intervention to improve symptom management in adults with long COVID: the COPE study protocol. Pilot Feasibility Stud. 2024 Jun 17;10(1):93. doi: 10.1186/s40814-024-01515-2. PMID 38886814